CLINICAL TRIAL: NCT04935385
Title: Monitoring Trace Element During Anesthesia Insertion and Surgery- A Prospective, Observational, Cohort Trial
Brief Title: Trace Element During Anesthesia Insertion and Surgery-
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0159-21
Record Dates: First submitted 2021-05-19; First posted 2021-06-23 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2021-05

CONDITIONS: Trace Elements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Following enrollment venous/ arterial blood samples will be collected from all study participants at the following timelines:
  1. At the beginning of surgery
  2. Following anesthesia induction prior to surgical site closure.
  3. At the end of surgery
  4. Additional blood sample will be drawn without inflicting pain to the patient 1 hour post surgery in some of the participants
  5. On the first day post-operatively, an additional sample may be collected for trace element analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: Patients aged 18 and above undergoing elective surgeries (including general surgery, neurosurgery, ear nose and throat surgeries, cardiac surgery, orthopedic surgeries, vascular surgeries and urological surgeries) at Rabin Medical Center under general anesthesia
  Interventions: Other: Collecting blood specimens

INTERVENTIONS:
Other: Collecting blood specimens — Blood samples will be collected from all study participants at different required timelines

SUMMARY:
Trace elements are micronutrients that are of vital important importance to human health and are involved in the process of many key human functions including the immune response, antioxidant defense and wound healing. Deficiency in a single element can manifest with multiple systems and can have significant organ impact.

Research has shown correlation between deficiencies in trace elements and increased risk for infections, sepsis, multi organ failure and mortality. However relatively few studies examined the impact of perioperative changes in trace elements and patients' postoperative outcomes.

In this prospective observational cohort study, we aim to examine the impact of perioperative changes in trace elements on postoperative outcomes, morbidity and mortality.

This study will include patients aged 18 and above undergoing elective surgeries under general anesthesia at Rabin Medical Center. In the operating room blood samples will be collected from all study participants in the beginning of surgery and at the end of surgery.

Collected samples will be sent for analysis of periodic table elements to assess the perioperative period changes in trace elements measured in whole blood. Participants intraoperative and postoperative data will be collected. All postoperative complications will be documented. Perioperative changes will be correlated with participants' postoperative outcomes using computer analytical correlations.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 and above
* Patients undergoing elective surgeries (as detailed above) under general anesthesia.
* Patients who can read and write Hebrew

Exclusion Criteria:

1. Emergency surgery
2. Regional anesthesia only

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 and above undergoing elective surgeries (including general surgery, neurosurgery, ear nose and throat surgeries, cardiac surgery, orthopedic surgeries, vascular surgeries and urological surgeries) at Rabin Medical Center under general anesthesia will be eligible for participation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-13 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
periodic trace elements measured in whole blood before and after surgery under general anesthesia. | 24 hours from surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center/Beilinson Campus, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided